CLINICAL TRIAL: NCT03861468
Title: Medico-economic and Quality of Life Evaluations in Obese Patients Followed by Medical Analysis Laboratories
Brief Title: Medico-economics and QoL of Obese Patients Followed by Medical Analysis Laboratories (BIOSAOS )
Acronym: BIOSAOS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Angers (Other Government); Poitiers University Hospital (Other); Union hospital, Toulouse (Unknown); Hospital Alpes Leman, Annemasse (Unknown); Hospital La Louvière, Lille (Unknown); Oriade Laboratory, Vizille (Unknown); Cerballiance laboratories, Lille (Unknown); Oriade laboratory, Annemasse (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 38RC17.360
Record Dates: First submitted 2019-02-22; First posted 2019-03-04 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Obesity Hypoventilation Syndrome; Obstructive Sleep Apnea
Keywords: obesity hypoventilation syndrome; obstructive sleep apnea; bicarbonates; STOP-BANG
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Sleep Apnea, Obstructive | interventions — Critical Pathways

STUDY DESIGN:
Intervention Model Description: Open, controlled, randomized clinical trial (cluster randomization)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Patients in the usual care group will be referred to their general practitioner (GP) / primary care practitioner as usual.
- Early care (Active Comparator): A different care pathway will be followed by the patients randomized to this group. They will be referred to a specialist (pneumologist) for OSA diagnosis and treatment if necessary
  Interventions: Other: Care pathway

INTERVENTIONS:
Other: Care pathway — Screening for OSA using a combination of bicarbonate assay and STOP-BANG questionnaire and further management by a pneumologist as necessary
  Arms: Early care

SUMMARY:
Obesity is a major risk factor for obstructive sleep apnea (OSA). However, OSA is still largely under diagnosed in patients with a high cardiovascular risk. In this population the STOP-BANG questionnaire facilitates OSA screening. Moreover, blood bicarbonate concentration is a simple tool to screen for chronic respiratory disease and if elevated, is a marker of cardiometabolic comorbidities in obese patients. A combination of blood bicarbonate concentration and STOP BANG score could provide a cost-effective method of screening for OSA in obese patients. Such screening could enable earlier management and might significantly reduce the costs of treatment and improve the quality of life of patients at 2 years.

DETAILED DESCRIPTION:
OSA is a frequent condition in the general population (3% of women and 10% of men), but remains largely undiagnosed. Obesity is a risk factor for OSA. Sleep apnea is associated with diurnal and nocturnal symptoms (snoring, somnolence, fatigue), and with increased cardiometabolic morbidity and mortality. Currently, continuous positive airway pressure (CPAP) is the gold-standard treatment for OSA and the cost-effectiveness of this treatment has already been demonstrated. Easy-to-use procedures to identify OSA patients earlier and thus to initiate treatment earlier, need to be developed and validated. The STOP-BANG questionnaire has been designed to facilitate the screening of OSA patients. Moreover, a measure of blood bicarbonate concentration is a simple method for screening for chronic respiratory diseases and a marker of cardiometabolic comorbidities. A combination of blood bicarbonate measurement and STOP-BANG score could permit earlier screening and less expensive care of obese patients. The hypothesize is that such OSA screening in the obese population (bicarbonates + STOPBANG) associated with earlier care (with treatment if necessary) could lead to improvement in quality of life of obese patients at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 80 years
* Obese (BMI ≥ 30kg/m²)
* Referred by GPs to the medical analysis laboratory for usual biological assessment
* Patients with no respiratory follow-up already in place
* Patient affiliated with a social protection plan
* Bicarbonate - Concentration ≥ 27 mmol/L
* STOP-BANG score ≥ 3
* Informed written consent signed by the patient

Exclusion Criteria:

* Acute disease or recently diagnosed chronic disease (< 2 months)
* Hospitalization for respiratory, metabolic or cardiovascular event (< 2 months)
* Renal insufficiency stage 4 or 5, or autoimmune disease, or viral hepatitis, or cirrhosis
* Cited persons in Sections L1121-5 to L1121-8 of the CSP (pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, a person who is the subject of a judicial or administrative legal protection)
* Patients already included in an interventional study (end of the study < 1 month)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
2-year medico-economic impact of the implementation of early care in obese patients with OSA | 24 months
  incremental cost-effectiveness ratio at 24 months calculated from the difference in healthcare costs between the 2 groups (early care vs usual care) adjusted to the difference in the number of quality adjusted life years

SECONDARY OUTCOMES:
Economic impact of the implementation of early care in obese patients with OSA over 3 years on the healthcare costs | 3 years
  The economic impact on healthcare costs from the Health Insurer's perspective will be calculated from the difference in healthcare costs between the two groups (early care vs usual care)
To evaluate the sensitivity of the screening tool | 24 months
  The sensitivity will be evaluated by comparison with polysomnography
To evaluate the specificity of the screening tool | 24 months
  The specificity will be evaluated by comparison with polysomnography
To evaluate the negative Predictive Value | 24 months
  The negative predictive value will be evaluated by comparison with polysomnography
To evaluate the positive predictive value of the screening tool | 24 months
  The positive predictive value will be evaluated by comparison with polysomnography
Clinical impact of the early care pathway on blood pressure at 12 months | 12 months
  Blood pressure at home
Clinical impact of the early care pathway on blood pressure at 24 months | 24 months
  Blood pressure at home
Clinical impact of the early care pathway on quality of life at 12 months | 12 months
  The EQ-5D-5L health status questionnaire, This scale is numbered from 0 to 100. 100 means the best health status. 0 means the worst health status.
Clinical impact of the early care pathway on quality of life at 24 months | 24 months
  The EQ-5D-5L health status questionnaire, This scale is numbered from 0 to 100. 100 means the best health status. 0 means the worst health status.
Clinical impact of the early care pathway (early care) on quality of life at 12 months | 12 months
  Stroke and Aphasia Quality of Life Scale (SAQOL), This questionnaire is intended to study the relationship between sleep and the quality of life. This scale is numbered from 0 to 4. higher values represent a worse outcome
Clinical impact of the early care pathway (early care) on quality of life at 24 months | 24 months
  Stroke and Aphasia Quality of Life Scale (SAQOL), This questionnaire is intended to study the relationship between sleep and the quality of life. This scale is numbered from 0 to 4. higher values represent a worse outcome
Clinical impact of the early care pathway on pharmacological treatments at 12 months | 12 months
  number of pharmacological treatments
Clinical impact of the early care pathway on pharmacological treatments at 24 months | 24 months
  number of pharmacological treatments
Impact on laboratory test results (troponin) at 12 months | 12 months
  troponin
Impact on laboratory test results (troponin) at 24 months | 24 months
  troponin
Impact on laboratory test results (NT-proBNP) at 12 months | 12 months
  NT-proBNP
Impact on laboratory test results (NT-proBNP) at 24 months | 24 months
  NT-proBNP
Impact on laboratory test results on cholesterol at 12 months | 12 months
  cholesterol
Impact on laboratory test results on cholesterol at 24 months | 24 months
  cholesterol
Impact on laboratory test results on triglycerides at 12 months | 12 months
  triglycerides
Impact on laboratory test results on triglycerides at 24 months | 24 months
  triglycerides
Impact on laboratory test results on glycaemia at 12 months | 12 months
  glycaemia
Impact on laboratory test results on glycaemia at 24 months | 24 months
  glycaemia
Impact on laboratory test results on Homeostasis model assessment (HOMA)-index at 12 months | 12 months
  Homeostasis model assessment (HOMA)-index
Impact on laboratory test results on Homeostasis model assessment (HOMA)-index at 24 months | 24 months
  Homeostasis model assessment (HOMA)-index
Impact on laboratory test results on hepatic transaminases at 12 months | 12 months
  transaminases (ASAT, ALAT)
Impact on laboratory test results on hepatic transaminases at 24 months | 24 months
  transaminases (ASAT, ALAT)
Impact on laboratory test results on creatinine at 12 months | 12 months
  creatinine
Impact on laboratory test results on creatinine at 24 months | 24 months
  creatinine
Impact on laboratory test results on C-Reactive Protein (CRP) at 12 months | 12 months
  C-Reactive Protein (CRP)
Impact on laboratory test results on C-Reactive Protein (CRP) at 24 months | 24 months
  C-Reactive Protein (CRP)
Impact on laboratory test results on alpha2-macroglobulin at 12 months | 12 months
  alpha2-macroglobulin
Impact on laboratory test results on alpha2-macroglobulin at 24 months | 24 months
  alpha2-macroglobulin

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, MD, PhD, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- ORIADE, Vizille, France

IPD SHARING:
Plan to Share IPD: Undecided